CLINICAL TRIAL: NCT00182455
Title: Topiramate Augmentation to a Selective Serotonin Re-uptake Inhibitor (SSRI) in Treatment-Resistant Generalized Social Phobia: A Double-Blind Placebo -Controlled Trial.
Brief Title: Efficacy of Adding Topiramate to Current Treatment in Treatment-Resistant Generalized Social Phobia (GSP)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: loss of funding
Sponsor: McMaster University (Other)
Collaborators: Janssen-Ortho Inc., Canada (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-080
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2018-04

CONDITIONS: Social Phobia
Keywords: Treatment Refractory Generalized Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Topiramate 25 - 400 mg/day x 12 weeks
  Interventions: Drug: Topiramate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — 25 - 400 mg/day x 12 weeks
  Other Names: Topomax
  Arms: 1
Drug: Placebo — 25 - 400 mg/day x 12 weeks
  Arms: 2

SUMMARY:
SSRI's are considered first-line treatments for GSP, however many patients continue to have significant symptoms despite an adequate trial of an SSRI. Topiramate, a drug, which targets the glutamate system in the brain, has been shown to improve symptoms of social phobia when used on its own and has also been used as an additive treatment in other anxiety disorders. This study will test the efficacy of adding topiramate to a subject's current SSRI in cases of GSP which are considered to be treatment-resistant.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with primary DSM-IV GSP
* Completion of an adequate trial (14 wks) of open, flexible dose SSRI treatment (fluoxetine 80mg/day, paroxetine 60mg/day, fluvoxamine 300 mg/day, sertraline 200mg/day, citalopram 60mg/day, escitalopram 30mg/day)
* Non or partial response to SSRI treatment (CGI-S > 4, LSAS > 40)

Exclusion Criteria:

* Any other DSM-IV Axis I primary diagnosis
* Meeting DSM-IV criteria for body dysmorphic disorder, eating disorder or current alcohol/substance abuse
* A lifetime history of bipolar affective disorder
* A Hx of schizophrenia/psychotic disorders, delirium, dementia, or amnestic/other cognitive disorders
* Borderline/antisocial personality disorder
* A comorbid Axis II cluster A personality disorder
* Hx of > 3 adequate trials with an SSRI
* score of > 4 on MADRS q.10
* Current increased risk of suicide
* Prior use of or an allergy to topiramate
* Participation in any clinical trial 30 days prior to entering the study
* Unable to tolerate being free of or shows signs of withdrawal benzodiazepines for 4 weeks
* Hx of seizures, kidney stones or thyroid problems
* BMI < 20

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression - Improvement (CGI-I) ≤ 2 | 12 weeks
Mean change in Liebowitz Social Anxiety Scale (LSAS) | 12 weeks

SECONDARY OUTCOMES:
Social Phobia Scale | 12 weeks
Social Phobia Inventory | 12 weeks
Clinical Global Impression -Severity | 12 weeks
Quality of life and Employment Satisfaction Questionnaire Sheehan Disability Scale | 12 weeks
Montgomery Asberg Depression Rating Scale | 12 weeks
Beck Depression Inventory | 12 weeks
Beck Anxiety Inventory | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada